CLINICAL TRIAL: NCT04125719
Title: A Phase IB Trial of PVSRIPO in Combination With Nivolumab in Patients With Recurrent PD-1 Refractory Melanoma
Brief Title: PVSRIPO in Combination With Nivolumab in Melanoma
Acronym: PPD1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: resubmission planned
Sponsor: Darell Bigner (Other)
Collaborators: Duke University (Other); Istari Oncology, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Darell Bigner, Edwin L. Jones, Jr. and Lucille Finch Jones Cancer Research Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00101803
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Primay PD-1 resistance (Experimental): Cohort 1 will include 15 patients who progressed within 3 months (primary resistance) of starting PD-1 therapy
  Interventions: Biological: PVSRIPO; Drug: Nivolumab
- Secondary PD-1 resistance (Experimental): Cohort 2 will include 15 patients who progressed after at least 3 months of PD-1 therapy
  Interventions: Biological: PVSRIPO; Drug: Nivolumab

INTERVENTIONS:
Biological: PVSRIPO — Intralesional injection of PVSRIPO
Drug: Nivolumab — Nivolumab infusion
  Other Names: Opdivo

SUMMARY:
In this study, patients with metastatic melanoma who have at least one injectable lesion that has been refractory to PD-1 therapy (n=30 patients) will be enrolled. Cohort 1 will include 15 patients who progressed within 3 months (primary resistance) of starting PD-1 therapy and cohort 2 will be patients who progressed after at least 3 months of PD-1 therapy. Patients will receive up to 7 injections of PVSRIPO intra-lesionally in combination with Nivolumab. Nivolumab will be administered according to the FDA-approved dosing schedule of 480 mg intravenously every 4 weeks, beginning ~10 days after the first PVSRIPO infusion and will continue for 4 cycles. Nivolumab may be continued up to 2 years per standard of care after the completion of the PVSRIPO injections.

DETAILED DESCRIPTION:
Patients must have histologically proven unresectable melanoma, stage IIIB, IIIC, IIID, or stage IV (AJCC staging must be documented in patient's medical record, as determined by CT of the chest, abdomen and pelvis, and/or whole body PET scan, and MRI of the brain within 4 weeks prior to administration of study drug). Patients must have failed PD-1 therapy as judged by the treating physician.

Patients will initially receive one injection of PVSRIPO intra-lesionally. Based on a phase 1 study of the agent in adult patients with recurrent GBM, the starting amount to be delivered will be 1x108 tissue culture infectious dose (TCID50) prior to initiation of nivolumab. Nivolumab will be administered according to the FDA-approved dosing schedule of 480 mg intravenously every 4 weeks, beginning ~10 days after the first PVSRIPO infusion and will continue for 4 cycles. PVSRIPO will then be given intralesionally to multiple lesions (if present) at days 38, 66, and 94.

At Day 108 after 4 doses of nivolumab and 4 treatments of PVSRIPO, imaging and a full disease assessment will be done and iRECIST determined. A patient with complete response (CR) or a partial response (PR) (at least at 75% decrease in the sum of all diameters of all target lesions plus new lesions) will continue on nivolumab for up to 2 years. For patients with PR (< 75% decrease), stable disease (SD), or progressive disease (PD), an additional 3 treatments of PVSRIPO q4weeks can be given concurrently with 3 doses of monthly nivolumab. The lesions will be chosen at discretion of principal investigator (PI) and can be new lesions, previously injected lesions, or untreated lesions. At Day 234 (±7 days), (after 7 total PVSRIPO injections and 8 doses of nivolumab), patients with PD will be off study, any patient with CR, PR, SD can receive up to 2 years total of nivolumab. If a patient has no remaining injectable lesions at any point during the study, PVSRIPO will not be given, but patients can continue on nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Positive serum anti-poliovirus antibody titer prior to biopsy.
2. The patient must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week prior to administration of the study agent.
3. Patient must have histologically proven unresectable melanoma, stage IIIB, IIIC, IIID, or stage IV (AJCC version 8 staging must be documented in patient's medical record, as determined by CT of the chest, abdomen and pelvis, and/or whole body PET scan, and MRI of the brain within 4 weeks prior to administration of study drug).
4. Patients must have progressed following ≥1 line of one prior systemic therapy, including immune checkpoint inhibitor (eg, anti- PD-1, ipilimumab, or anti PD-1 plus ipilimumab); and if BRAF V600 mutation-positive, after a BRAF inhibitor or BRAF inhibitor in combination with MEK inhibitor. Patients last dose of systemic therapy must have been within 9 months prior to signing consent for this study. Patients treated in the adjuvant setting and develop recurrence are also allowed.
5. Cohort 1 will include 15 patients who progressed within 3 months (primary resistance) of starting PD-1 therapy and cohort 2 will be patients who progressed after at least 3 months of PD-1 therapy.
6. Patient must be ≥18 years of age.
7. Patient must have an ECOG/Zubrod status of 0-1.
8. Patient's disease must be bi-dimensionally measurable by caliper or radiological method as defined in the iRECIST criteria. The sum of target lesion diameters should be at least 10 mm.
9. At least 1 injectable cutaneous, subcutaneous or nodal melanoma lesion ≥ 10 mm in longest diameter or, multiple injectable melanoma lesions which in aggregate have a longest diameter of ≥ 10 mm.
10. Serum lactate dehydrogenase (LDH) levels less than 1.5 x upper limit of normal (ULN).
11. Patient must have adequate bone marrow, liver and renal function as assessed by the following:

    1. Hemoglobin ≥ 9.0 g/dl, patients may be transfused to meet this criteria
    2. Lymphocyte count ≥ 0.5 x 109/L (500 µL)
    3. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500 µL)
    4. Platelet count ≥ 100 x 109/L (100,000 µL) without transfusion
    5. AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions:

    i. Patients with documented liver metastases: AST and ALT ≤ 5 x ULN ii. Patients with documented liver or bone metastases: ALP ≤ 5 x ULN f. Serum bilirubin ≤ 1.5 x ULN with the following exception: i. Patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN g. Serum creatinine ≤ 1.5 x ULN h. Serum albumin ≥ 25 g/L (2.5 g/dL) i. For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN
12. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
13. Patients must have a life expectancy of > 6 months.
14. Patient must provide a signed and dated written informed consent prior to registration and any study-related procedures.
15. Ability to read and understand English and the ability to complete paper and electronic survey assessments.
16. Ability to comply with the study protocol, in the investigator's judgement.
17. For women of childbearing potential:

    1. Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the last dose of study treatment. Note: A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

    i. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

    ii. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
18. For men:

    a. Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: i. With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 7 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

ii. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Symptomatic, untreated, or actively progressing CNS metastases. Patients with a history of treated CNS lesions are eligible, provided that all of the following criteria are met:

   1. The patient has not received stereotactic radiotherapy within 7 days prior to initiation of study treatment or whole-brain radiotherapy within 14 days prior to initiation of study treatment.
   2. The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.
   3. Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
2. History of leptomeningeal disease.
3. Uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at study entry.

   1. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
   2. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

   a. Patients with indwelling catheters (e.g., PleurX®) are allowed.
5. Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN).
6. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   i. Rash must cover < 10% of body surface area ii. Disease is well-controlled at baseline and requires only low-potency topical corticosteroids iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
7. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

   a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
8. History of a Positive HIV test
9. Known active hepatitis B virus (HBV) infection (chronic or acute).

   a. Patients who have had a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test are eligible for the study.
10. Known active hepatitis C virus (HCV) infection.

    a. If potential subjects have a history of a positive HCV antibody test, but negative HCV RNA test, subject may be eligible for the study
11. Active tuberculosis
12. Significant cardiovascular disease, such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
13. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study.
14. History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
15. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
16. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment (note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study).
17. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
18. Prior allogeneic stem cell or solid organ transplantation.
19. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study or within 5 months after the last dose of nivolumab.
20. Treatment with investigational therapy within 15 days prior to initiation of study treatment
21. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment.
22. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

    1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator approval has been obtained. However, during the course of the study, use of corticosteroids is allowed if used for treating irAEs, adrenal insufficiencies, or if administered at doses of prednisone ≤ 10 mg daily or equivalent.
    2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
23. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
24. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the nivolumab formulation.
25. Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the last dose of study treatment.
26. Women of childbearing potential must have a negative serum pregnancy test result within 24 hours prior to the initial administration of the study drug and then every 4 weeks during the treatment period.
27. Patients with human serum albumin allergy.
28. Patients with a previous history of neurological complications due to PV infection.
29. Patients with a history of prior serious immune related adverse events while receiving PD-1 therapy.
30. Patients with undetectable anti-tetanus toxoid IgG
31. Patients with known history of agammaglobulinemia
32. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups.
33. Prior allogeneic stem cell transplantation
34. Psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance; any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of Nivolumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea
35. Prisoners, or subjects who are compulsory detained.
36. Inablility to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Assess the percent of adverse events related to the combination of PVSRIPO + nivolumab in the treatment of patients with recurrent melanoma. | 36 months
  Toxicities will be measured based on the number of adverse events as measured by clinical exams.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Beasley, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No